CLINICAL TRIAL: NCT07046403
Title: A Multicentric Randomized Controlled Clinical Trial Comparing the Use of High Purity Type-I Collagen-Based Skin Substitute vs. Dehydrated Human Amnion/Chorion Membrane in the Treatment of Diabetic Foot Ulcers
Brief Title: Multicentric RCT Comparing High Purity Type I Collagen-Skin Substitute vs dHACM in Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adichunchanagiri Institute of Medical Sciences, B G Nagara (Other)
Collaborators: Mysore Medical College and Research Institute (Other); Rajarajeswari Dental College & Hospital (Other); JSS Medical College Hospital (Unknown)
Responsible Party: Principal Investigator, Dr Naveen Narayan MS, MCh (Plastic Surgery), Professor & HoD, Department of Plastic Reconstructive & Aesthetic Surgery, Adichunchanagiri Institute of Medical Sciences, B G Nagara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIMS/IEC/206/2025
Record Dates: First submitted 2025-06-21; First posted 2025-07-01 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Ulcer (DFU)
Keywords: Diabetic Foot Ulcer; High Purity Type-I Collagen-Based Skin Substitute; Dehydrated Human Amnion/Chorion Membrane; Randomized Controlled Clinical Trial; Multicentric Study
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High Purity Type-I Collagen-based Skin Substitute and SOC (Active Comparator): The SOC in this study is wound care covering with High Purity Type-I Collagen-based Skin Substitute applied weekly or as needed followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous paraffin gauze (Cuticel), second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap (Crepe Bandage)
  Interventions: Device: High Purity Type-I Collagen-based Skin Substitute and SOC
- Human Amnion/Chorion Membrane and SOC (Active Comparator): The SOC in this study is wound care covering with Dehydrated Human Amnion/Chorion Membrane followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous paraffin gauze (Cuticel), second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap (Crepe Bandage)
  Interventions: Device: Dehydrated Human Amnion / Chorion Membrane and SOC

INTERVENTIONS:
Device: High Purity Type-I Collagen-based Skin Substitute and SOC — The SOC in this study is wound care covering with High Purity Type-I Collagen-based Skin Substitute applied weekly or as needed followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous paraffin gauze (Cuticel), second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap (Crepe Bandage)
  Arms: High Purity Type-I Collagen-based Skin Substitute and SOC
Device: Dehydrated Human Amnion / Chorion Membrane and SOC — The SOC in this study is wound care covering with Dehydrated Human Amnion/Chorion Membrane followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous paraffin gauze (Cuticel), second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap (Crepe Bandage)
  Arms: Human Amnion/Chorion Membrane and SOC

SUMMARY:
This is a randomized controlled clinical investigation in patients suffering from diabetic foot ulcers at multiple centers. The study intends to compare patient outcome data using Standard of Care with Type-I Collagen-based Skin Substitute and Standard of Care with Dehydrated Human Amnion/Chorion Membrane.

DETAILED DESCRIPTION:
The purpose of the present study is to compare the safety and efficacy of high-purity type-I collagen-based skin substitutes (HPTC), which are free from contaminants such as lipids, elastin, and other immunogenic particles, versus dehydrated human amnion/chorion membrane (dHACM) in the treatment of DFUs. This multicentric randomized, controlled clinical trial seeks to provide valuable insights into the best treatment strategy for enhancing healing outcomes and reducing the challenges posed by chronic DFUs.

Study will be carried out as a multicentric randomized, controlled open-label study to evaluate the safety and effectiveness of High Purity Type-I Collagen-based Skin Substitute (HPTC) compared to Dehydrated Human Amnion/Chorion Membrane (dHACM) for treating diabetic foot ulcers (DFUs). The trial will include patients with DFUs treated by wound care specialists at Adichunchanagiri Institute of Medical Sciences (AIMS), B. G. Nagara, Rajarajeswari Medical College and Hospital (RRMCH), Bangalore, JSS Medical College and Hospital (JSS), Mysore and Mysore Medical College and Research Institute (MMC&RI), Mysore, under the supervision of primary investigator Dr Naveen N. the other principal investigators include Dr Kamal Kumar M, Dr Ravi Shivaiah and Dr Vijay Kumar, respectively. Informed consent will be obtained from all participants prior to any study-related procedures at each of the 3 centres. Each patient will sign an Institutional Ethics Committee / Investigational Review Board (IEC/IRB)-approved consent form, at respective participating centres. IEC/IRB of Adichunchanagiri Institute of Medical Sciences, B. G. Nagara, will be the Designated Ethics Committee (DEC).

The study population will consist of patients seeking treatment for DFUs. Eligible patients will be those willing to participate and comply with scheduled visits on days 7, 10, 14, 17, 21, and 28. The study will include two phases: screening and treatment.

The screening phase aimed to determine patient eligibility for the treatment phase.

Centralized computer-generated block randomization, stratified by centre in a 1:1 ratio will be done. Due to the nature of the interventions, blinding of participants and clinicians is not feasible. However, outcome assessors and data analysts will be blinded to treatment allocation to minimize bias.

The treatment phase of the study will commence with a series of evaluations to ensure patients remained eligible. Participants who will continue to meet the inclusion criteria after the screening phase will be randomly assigned to one of two groups:

1. Standard of Care (SOC) with High Purity Type-I Collagen-based Skin Substitute (HPTC).
2. Standard of Care (SOC) with Dehydrated Human Amnion/Chorion Membrane (dHACM). Neither the patients nor the clinicians will be blinded to group assignments. The randomization will follow a balanced schedule, using permuted blocks of 12. When a patient will be ready for randomization, the study site will contact a representative from the sponsor, who will open a sequentially numbered opaque envelope to disclose the group assignment, maintaining allocation concealment.

Throughout the 4-week treatment phase, patients will be reassessed on days 7, 10, 14, 17, 21, and 28. The SOC dressing applied in both groups consisted of a three-layer system:

* First layer: Non-adherent, porous paraffin gauze.
* Second layer: Absorbent gauze pads.
* Third layer: Soft roll and Crepe bandage. If the study ulcer was found to be 100% re-epithelialized during the visit, no further study procedures will be conducted at that time. The patient will then be scheduled for a follow-up visit after one week to confirm the healing.

If full healing was not achieved, an evaluation will be carried out to check for any signs of clinical infection. If an infection is confirmed, treatment with topical antimicrobials or oral antibiotics will be permitted, though the use of topical antibiotics will be prohibited.

After this infection assessment, the ulcer would be cleaned, photographed, and debrided at the investigator's discretion to ensure a clean and granulating wound base with minimal adherent slough. The Standard of Care (SOC) will be then re-applied, and patients will be instructed to keep the bandage dry. Additionally, they will be advised to contact or return to the study site if the bandage became soiled or removed.

Study Completion Patients will complete the study 4 weeks after their initial treatment visit. However, if a patient's study ulcer healed before the 4-week period, they will be considered to have completed the study at the time of full healing.

Complete healing will be defined as 100% re-epithelialization of the ulcer with no drainage. Throughout the study, patients will retain the right to decline participation or withdraw at any time without prejudice.

In the event of a patient's withdrawal, their last recorded wound measurement will be carried forward to determine the change in wound size and calculate their final outcome.

Study Outcomes

Primary Endpoint:

• The primary outcome of the study will be the proportion of subjects who achieved improvement in wound healing, as observed on days 7, 10, 14, 17, 21, and 28. The wound closure of the target ulcer will be continuously monitored until the end of the 4-week period.

Secondary Endpoints:

* Vascular Incursion: To assess the infiltration of vascularity in the ulcer bed on day 5 post-treatment initiation (using HPE analysis by taking 2 mm diameter punch biopsy samples).
* Time to Achieve Complete Wound Closure: Time taken for the target ulcer to achieve complete wound closure will be assessed on days 7, 10, 14, 17, 21, and 28.
* Percentage Wound Area Reduction: This will be measured weekly on days 7, 10, 14, 17, 21, and 28 using digital photography.
* Mean Number of Repeated Applications of HPTC: The average number of times the reapplication of High Purity Type-I Collagen-based Skin Substitute (HPTC) to achieve wound closure will be documented as part of the study process.
* To monitor incidence of infection or complications
* To assess patient-reported quality of life
* To evaluate scar quality using validated scales (e.g., Vancouver Scar Scale)

Exploratory Endpoint:

• The appearance, structural stability, and fragility of the newly formed skin will be documented at each visit. Any recurrence of the wound will also be monitored.

Statistical Analysis

Data will be analysed on an intention-to-treat basis. Continuous variables will be summarized using means and standard deviations or medians and interquartile ranges, as appropriate. Categorical variables will be presented as frequencies and percentages. Comparative analyses will include:

* Descriptive statistics for baseline characteristics
* Chi-square tests for categorical outcomes.
* Independent t-tests or Mann-Whitney U tests for continuous outcomes.
* Kaplan-Meier survival analysis for time-to-event data, with log-rank tests to compare groups.

Multivariable regression models will adjust for potential confounders, such as baseline wound size and patient comorbidities.

Sample Size Calculation Based on previous studies, assuming a 20% difference in the primary outcome between groups, with 60% healing in the dHACM group and 80% in the HPTC group, a sample size of 60 participants per group (total N=60) combined from the 4 centres will provide 80% power to detect this difference at a 5% significance level, accounting for a 10% dropout rate.

Ethical Considerations The study will adhere to the Declaration of Helsinki principles and Good Clinical Practice guidelines. Ethical approval will be obtained from Institutional Ethics Committee of all participating centres. Informed consent will be obtained from all participants before enrolment. Adverse events will be monitored and reported. Participant confidentiality will be maintained, and data will be anonymized. Findings will be submitted to peer-reviewed journals and presented at relevant conferences.

Timeline Recruitment: 1 month Intervention & follow-up assessment: 3 months Data analysis and reporting: 1 month

Potential Implications This study aims to provide robust evidence on the comparative efficacy of HPTC and dHACM in managing DFUs. If HPTC proves superior to dHACM alone, it could establish a standard in treating DFUs, reducing healing time. Positive findings could influence clinical practice guidelines, offering alternative treatment options that may enhance patient outcomes and reduce healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age or older.
* Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
* At randomization subjects must have a target diabetic foot ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 10.0 cm2 measured post debridement using a ruler to measure wound area.
* The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
* The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
* The target ulcer must be full thickness on the foot or ankle that does not probe to bone.
* Adequate circulation to the affected foot as documented by any of the following methods performed within 3 months of the first screening visit:

Transcutaneous Oxygen Measurement (TCOM) ≥30 mmHg Ankle-Brachial Index (ABI) between 0.7 and 1.3 Peripheral Vascular Resistance (PVR): Biphasic Toe-Brachial Index (TBI) ˃0.6 As an alternative, arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle of the target extremity.

* If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
* The subject must consent to using the prescribed off-loading method for the duration of the study.
* The subject must agree to attend the twice-weekly/weekly study visits required by the protocol.
* The subject must be willing and able to participate in the informed consent process.
* Patients must have read and signed the IRB approved ICF before screening procedures are undertaken.

Exclusion Criteria:

* A subject known to have a life expectancy of <6 months.
* If the target ulcer is infected or if there is cellulitis in the surrounding skin.
* Presence of osteomyelitis or exposed bone, probes to bone or joint capsule on investigator's exam or radiographic evidence.
* A subject that has an infection in the target ulcer that requires systemic antibiotic therapy.
* A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy.
* Topical application of steroids to the ulcer surface within one month of initial screening.
* A subject with a previous partial amputation on the affected foot is excluded if the resulting deformity impedes proper offloading of the target ulcer.
* A subject with a glycated hemoglobin (HbA1c) greater than or equal to 13% taken at or within 3 months of the initial screening visit.
* A subject with a serum creatinine ≥ 3.0mg/dL within 6 months of the initial screening visit.
* A subject with an acute Charcot foot, or an inactive Charcot foot, that impedes proper offloading of the target ulcer.
* Women who are pregnant or considering becoming pregnant within the next 6 months.
* A subject with end stage renal disease requiring dialysis.
* A subject who participated in a clinical trial involving treatment with an investigational product within the previous 30 days.
* A subject who, in the opinion of the Investigator, has a medical or psychological condition that may interfere with study assessments.
* A subject treated with hyperbaric oxygen therapy or a Cellular and/or Tissue Product (CTP) in the 30 days prior to the initial screening visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-07-05 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prema Dhanraj, MS, MCh, Study Chair — Rajarajeshwari Medical College and Hospital
Locations (4):
- India (4):
  - RajaRajeswari Medical College and Hospital, Bangalore, Karnataka
  - Adichunchanagiri Institute of Medical Sciences, Mandya, Karnataka
  - Mysore Medical College and Research Institute, Mysore, Karnataka
  - JSS Medical College Hospital, Mysore, Karnataka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Narayan N, Gowda S, Shivannaiah C. A Randomized Controlled Clinical Trial Comparing the Use of High Purity Type-I Collagen-Based Skin Substitute vs. Dehydrated Human Amnion/Chorion Membrane in the Treatment of Diabetic Foot Ulcers. Cureus. 2024 Dec 5;16(12):e75182. doi: 10.7759/cureus.75182. eCollection 2024 Dec. PMID 39649230
- [Background] Wolfe EM, Mathis SA, de la Olivo Munoz N, Ovadia SA, Panthaki ZJ. Comparison of human amniotic membrane and collagen nerve wraps around sciatic nerve reverse autografts in a rat model. Biomater Biosyst. 2022 Apr 7;6:100048. doi: 10.1016/j.bbiosy.2022.100048. eCollection 2022 Jun. PMID 36824162
- [Background] Mohammed YA, Farouk HK, Gbreel MI, Ali AM, Salah AA, Nourelden AZ, Gawad MMA. Human amniotic membrane products for patients with diabetic foot ulcers. do they help? a systematic review and meta-analysis. J Foot Ankle Res. 2022 Sep 14;15(1):71. doi: 10.1186/s13047-022-00575-y. PMID 36104736
- [Background] DiDomenico LA, Orgill DP, Galiano RD, Serena TE, Carter MJ, Kaufman JP, Young NJ, Jacobs AM, Zelen CM. Use of an aseptically processed, dehydrated human amnion and chorion membrane improves likelihood and rate of healing in chronic diabetic foot ulcers: A prospective, randomised, multi-centre clinical trial in 80 patients. Int Wound J. 2018 Dec;15(6):950-957. doi: 10.1111/iwj.12954. Epub 2018 Jul 17. PMID 30019528
- [Background] Huang Y, Kyriakides TR. The role of extracellular matrix in the pathophysiology of diabetic wounds. Matrix Biol Plus. 2020 Apr 22;6-7:100037. doi: 10.1016/j.mbplus.2020.100037. eCollection 2020 May. PMID 33543031
- [Background] Singh N, Armstrong DG, Lipsky BA. Preventing foot ulcers in patients with diabetes. JAMA. 2005 Jan 12;293(2):217-28. doi: 10.1001/jama.293.2.217. PMID 15644549
- [Background] Narayan N, Shivannaiah C, Gowda S. Evaluating the Efficacy of High-Purity Type I Collagen-Based Skin Substitute Versus Dehydrated Human Amnion/Chorion Membrane in the Treatment of Venous Leg Ulcers: A Randomized Controlled Clinical Trial. Cureus. 2025 Jul 30;17(7):e89031. doi: 10.7759/cureus.89031. eCollection 2025 Jul. PMID 40747200
- [Background] Narayan N, Ramegowda YH, Raghupathi DS, Chethan S, Gowda S. Biological Skin Substitutes in Pressure Ulcers: High-Purity Type I Collagen-Based Versus Amnion/Chorion Membrane. Cureus. 2025 Aug 25;17(8):e90956. doi: 10.7759/cureus.90956. eCollection 2025 Aug. PMID 40862036

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (8.2) | 53.1 (9.1) | 52.75 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 42 | 38 | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 60 | 60 | 120
BMI (kg/m²) [Mean (Standard Deviation); unit: kg/m^2] | 26.8 (3.4) | 26.2 (3.8) | 26.5 (3.6)
Diabetes duration (years) [Mean (Standard Deviation); unit: years] | 12.6 (5.8) | 13.2 (6.4) | 12.9 (6.1)
HbA1c (as percentage) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.4 (1.6) | 8.7 (1.8) | 8.6 (1.7)
Ulcer duration (weeks) [Mean (Standard Deviation); unit: weeks] | 8.4 (4.2) | 8.9 (4.6) | 8.7 (4.4)
Ulcer size (cm²) [Mean (Standard Deviation); unit: square centimeters] | 10.4 (3.2) | 9.8 (2.9) | 10.1 (3.1)
Ankle-Brachial Index (ABI) [Mean (Standard Deviation); unit: ratio] — A normal ABI is between 1.0 and 1.4, while a score below 0.9 can indicate peripheral arterial disease (PAD).
  1. Borderline: 0.91 to 0.99
  2. Mild to moderate PAD: 0.41 to 0.90
  3. Severe PAD: 0.40 or less
  4. Higher scores above 1.4 may suggest that the arteries are stiff and not compressible such as in Diabetes Mellitus.
  How to calculate - The blood pressure is measured in an artery in each arm. The blood pressure is measured in an artery in each ankle. The higher systolic blood pressure from the ankle is divided by the higher systolic blood pressure from the arm to get the ABI.
  ratio | 0.94 (0.18) | 0.91 (0.16) | 0.93 (0.17)
Previous ulcer history [Count of Participants; unit: Participants] | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Wound Area
Description: The primary outcome of the study will be the percentage change in wound area, assessed at 1, 2,3, and 4 weeks, and week 5 reported measured manually with digital photography.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
Number analyzed (Participants) | 60 | 60
percentage change | 81.5 (12.3) | 64.2 (14.1)

2. Secondary Outcome: Histopathological Analysis
Description: Histopathological assessment will be done using biopsy on Day 0 of application to be compared with Day 5 after application of Type-I Collagen-based Skin Substitute or Human Amnion/Chorion Membrane. Histopathology assessed at day 0 and day 5, day 5 reported. Subsequently histopathology of biopsy will be done to look for:
  vascular infiltration (0-3 scale) - higher score means better, neo-epithelialization (0-3 scale) - higher score means better, fibroblast activity (0-3 scale) - higher score means better, inflammatory response (0-3 scale) - lower score means better and collagen deposition (0-3 scale) - higher score means better
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
Number analyzed (Participants) | 60 | 60
score on a scale
  vascular infiltration (0-3 scale) | 2.4 (0.6) | 1.8 (0.7)
  neo-epithelialization (0-3 scale) | 2.6 (0.5) | 2.1 (0.6)
  fibroblast activity (0-3 scale) | 2.5 (0.6) | 1.9 (0.7)
  inflammatory response (0-3 scale) | 1.2 (0.4) | 1.8 (0.6)
  collagen deposition (0-3 scale) | 2.3 (0.7) | 1.7 (0.8)

3. Secondary Outcome: Histopathological Analysis - Capillary Density (Vessels Per mm²)
Description: Histopathological assessment will be done using biopsy on Day 0 of application to be compared with Day 5 after application of Type-I Collagen-based Skin Substitute or Human Amnion/Chorion Membrane. Histopathology assessed at day 0 and day 5, day 5 reported. Subsequently histopathology of biopsy will be done to look for capillary density (vessels per mm²) - higher count means better
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: vessels per mm²
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
Number analyzed (Participants) | 60 | 60
vessels per mm² | 45.6 (7.9) | 29.4 (9.2)

4. Secondary Outcome: Percentage of Participants to Obtain Complete Wound Closure
Description: The percentage of participants that obtain complete wound closure over the 5 weeks (4 weeks treatment period plus 1 week follow up)
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
Number analyzed (Participants) | 60 | 60
Participants | 50 | 31

5. Secondary Outcome: Time to Achieve Complete Wound Closure
Description: Complete wound closure is defined as full epithelialization of the wound with no need for dressings, and sustained closure without signs of infection or breakdown.Time taken for the target ulcer to achieve this will be assessed on days 7, 14, 21, 28 and 35.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
Number analyzed (Participants) | 60 | 60
days | 22.2 (5.4) | 28.8 (6.2)

6. Secondary Outcome: Percentage of Participants Achieving ≥50% Wound Healing
Description: Measurement of percentage of participants achieving ≥50% wound healing (epithelialization) assessed at follow up
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
Number analyzed (Participants) | 60 | 60
Participants | 53 | 33

7. Secondary Outcome: Mean Number of Applications of HPTC / dHACM
Description: The average number of applications of High Purity Type-I Collagen-based Skin Substitute (HPTC) or dehydrated human amniotic/chorionic membrane (dHACM) to achieve wound closure will be documented as part of the study process.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: number of applications
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
Number analyzed (Participants) | 60 | 60
number of applications | 2.8 (1.2) | 3.4 (1.6)

8. Secondary Outcome: Number of Participants With Adverse Events
Description: To monitor number of participants with adverse events related to the intervention (e.g., infection, allergic reactions)
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
Number analyzed (Participants) | 60 | 60
Participants | 4 | 11

9. Secondary Outcome: Patient-Reported Quality of Life Assessed Using Diabetic Foot Ulcer Scale - Short Form (DFS-SF)
Description: The Diabetic Foot Ulcer Scale - Short Form (DFS-SF) is a validated, disease-specific health-related quality of life (HRQoL) questionnaire designed to assess the impact of diabetic foot ulcers on patients' wellbeing evaluating four validated sub-scales:
  Physical Functioning Daily Activities Emotions Social Functioning
  Subscale Scoring: Scores range from 0-100 for each sub-scale, with higher scores indicating better quality of life. Data were collected at baseline and at Weeks 2, 4, and 5, and week 5 results reported
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale (0-100)
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
Number analyzed (Participants) | 60 | 60
Scores on a scale (0-100)
  Physical functioning | 78.6 (14.2) | 68.4 (16.8)
  Daily activities | 76.2 (13.6) | 62.8 (15.4)
  Emotions | 82.4 (12.8) | 71.6 (16.2)
  Social functioning | 79.8 (15.2) | 65.2 (17.6)

10. Secondary Outcome: Healed Wound Appearance Assessment Using Vancouver Scar Scale
Description: The resultant new skin is assessed and documented at each visit up to 5 weeks and week 5 visit reported using the Vancouver Scar Scale assessing vascularity, pigmentation, pliability and height/thickness with total score ranging from 0 to 13 (lesser the score better the scar)
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale (0-13)
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
Number analyzed (Participants) | 60 | 60
scores on a scale (0-13) | 4.2 (2.1) | 6.8 (2.8)

ADVERSE EVENTS:
Time Frame: 5 weeks - From first application (Week 0) through end of follow-up (Week 5).
Description: All the study participants were considered at risk for adverse events.
Arm/Group | High Purity Type-I Collagen-based Skin Substitute and SOC | Human Amnion/Chorion Membrane and SOC
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 4/60 | 11/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Purity Type-I Collagen-based Skin Substitute and SOC (N=60) | Human Amnion/Chorion Membrane and SOC (N=60)
Local irritation (Skin and subcutaneous tissue disorders) | 1 | 3
Minor allergy (Skin and subcutaneous tissue disorders) | 1 | 4
Mild infection (Skin and subcutaneous tissue disorders) | 2 | 4

LIMITATIONS AND CAVEATS:
The study utilized an open-label design, which may introduce performance and detection bias. The follow-up duration of 5 weeks was predetermined and may not allow full evaluation of long-term wound durability or recurrence. The study did not include a pre-planned economic or cost-effectiveness assessment. The study was conducted at selected clinical sites and enrolled a specific diabetic population as per the inclusion/exclusion criteria, which may restrict broader applicability of findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT07046403/Prot_SAP_001.pdf